CLINICAL TRIAL: NCT05049655
Title: Multi-Center Clinical Database of Infants for the Investigation of Early Nutrition Biomarkers
Status: Enrolling by invitation | Type: Observational
Sponsor: ByHeart (Industry)
Responsible Party: Sponsor
Other Study IDs: BH-10118-02
Record Dates: First submitted 2021-09-09; First posted 2021-09-20 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Infant Development

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Cohort 1: Babies who were fed commercial formula, study formula, or were fed with human milk in the SS-101-18 study that consented to the BH-10118-02 study
- Cohort 2: Babies fed with commercial formula (including ByHeart formula) or fed with human milk

SUMMARY:
An observational study to generate a long-term outcome database from medical records for infants who completed protocol SS-101-18 or infants who are breastfed, fed commercial formula, or fed a marketed ByHeart formula.

DETAILED DESCRIPTION:
The first Cohort (Cohort 1) goals of the registry include: to compile a clinical database of children who were fed in SS-101-18 by breastfeeding, commercial formula, or ByHeart formula; to investigate any difference in demographics, growth, development, medical diagnoses, and outcomes between the feeding groups, and in particular to compare ByHeart formula-fed infants against commercial formula-fed infants, and referenced against breastfed infants.

The second Cohort (Cohort 2) goals of the registry include: to compile a clinical database of children who were fed by breastfeeding or commercial formula (including ByHeart formula); to describe any difference in growth, development, medical diagnoses, and outcomes based on early nutritional intake; and to inform or facilitate development of future ByHeart products.

ELIGIBILITY:
Inclusion Criteria Cohort 1:

* Active participation in SS-101-18 through Visit 9
* Provision of signed and dated informed consent form (ICF) by parent or legally authorized representative (LAR)
* Stated willingness to comply with all study procedures by parent or LAR.

Exclusion Criteria Cohort 1:

* Did not participate in SS-101-18
* Participated in SS-101-18 that withdrew from the study for any reason prior to Visit 9
* Anything that in the opinion of the Investigator is likely to interfere with participation in the registry.

Inclusion Criteria Cohort 2:

* Be less than 120 days old at the time of enrollment
* Provision of signed and dated informed consent form (ICF) by parent or legally authorized representative (LAR)
* Stated willingness to comply with all study procedures by parent or LAR.

Exclusion Criteria Cohort 2:

* Participation in SS-101-18
* Anything that, in the opinion of the Investigator, is likely to interfere with participation in the registry.
* In the opinion of the investigator, has a diagnosed medical condition or genetic abnormality known to impact growth or development.

Ages: 0 Days to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Approximately 2000 infants will be enrolled in this study.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2021-10-19 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Cohort 1: Growth, Development, Diagnoses, and Long-term Outcomes | 5 years
  The registry will be utilized to investigate growth, development, diagnoses, and long-term outcomes of infants who received ByHeart study formula, commercially available formula, or breastmilk in the SS-101-18 protocol.
Cohort 2: Growth, Development, Diagnoses, and Long-term Outcomes | 5 years
  A clinical database of children of all feeding options; to describe any difference in growth, development, medical diagnoses, and outcomes based on early nutritional intake

CONTACTS AND LOCATIONS:
Overall Officials: Devon Kuehn, M.D., Study Director — ByHeart
Locations (9):
- United States (9):
  - Alabama Clinical Therapeutics, LLC (Cohort 1), Birmingham, Alabama
  - Watching Over Mothers & Babies (Cohort 1), Tuscan, Arizona
  - The Children's Clinic of Jonesboro (Cohort 1), Jonesboro, Arkansas
  - Clinical Research Prime (Cohort 1), Idaho Falls, Idaho
  - Pediatric Associates Mt. Carmel (Cohort 1), Cincinnati, Ohio
  - Coastal Pediatric Research (Cohort 1), Charleston, South Carolina
  - Coastal Pediatric Research (Cohort 1), Summerville, South Carolina
  - Holston Medical Group (Cohort 1), Kingsport, Tennessee
  - Tanner Clinic (Cohort 1), Layton, Utah

IPD SHARING:
Plan to Share IPD: Undecided